CLINICAL TRIAL: NCT02810756
Title: Proof of Principle and Pharmacological Phase 0 Study With Improved Solubility Pazopanib
Brief Title: Study With Improved Solubility Pazopanib
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N16PZN
Record Dates: First submitted 2016-05-31; First posted 2016-06-23 (Estimated); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Pharmacokinetics of Pazopanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treated patients (Experimental)
  Interventions: Drug: New Pazopanib formulation

INTERVENTIONS:
Drug: New Pazopanib formulation

SUMMARY:
The pharmacokinetics of a new formulation with Pazopanib will be studied. This will be done in a patient cohort of n = 12.

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced or metastatic cancer;
* Able and willing to give written consent;
* WHO performance status of 0, 1 or 2;
* Able and willing to undergo blood sampling for PK analysis;
* Minimal acceptable safety laboratory values;
* Negative pregnancy test for female patients with childbearing potential;
* Able and willing to swallow oral medication.

Exclusion Criteria:

* Any treatment with investigational drugs within 30 days prior to receiving the investigational treatment;
* Any treatment with CYP3A4, BCRP or PGP interfering drugs;
* Patients who received treatment with Votrient(R) kess than 1 week ago;
* Woman who are pregnant or breast feeding;
* Patients suffering from any known condition that may influence the dissolution or absorption of Pazopanib.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-09-15 (Actual); Primary Completion 2017-08-28 (Actual); Study Completion 2017-08-28 (Actual)

PRIMARY OUTCOMES:
Plasma concentration | 24 hours
  Concentration of pazopanib in plasma

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 1 week
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0
Area under the plasma concentration versus time curve (AUC) | 24 hours
  Area under the plasma concentration versus time curve (AUC)

CONTACTS AND LOCATIONS:
Locations (1):
- Netherlands Cancer Institute, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No
Individual participant data will remain confidential